CLINICAL TRIAL: NCT02308787
Title: Multicenter, Retrospective Data Collection of Routine Clinical Use With the Spectra Optia® Apheresis System for Platelet Depletion Procedures.
Brief Title: Retrospective Data Collection of Routine Use With Spectra Optia® for Platelet Depletions
Acronym: PLTD
Status: Completed | Type: Observational
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Other Study IDs: CTS-5052
Record Dates: First submitted 2014-11-18; First posted 2014-12-04 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Thrombocythemia; Myeloproliferative Disease; Thrombocytosis
Keywords: platelet depletion; apheresis
MeSH Terms: conditions — Thrombocytosis; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Spectra Optia Apheresis System — Platelet Depletion

SUMMARY:
Multicenter, Retrospective Data Collection of Routine Clinical Use with the Spectra Optia® Apheresis System for Platelet Depletion Procedures.

DETAILED DESCRIPTION:
This is a multicenter, retrospective data collection to evaluate the in routine use performance and safety of platelet depletions performed via the Spectra Optia system. Data collection will include procedures in 2- 3 different centers in Europe done between November 2011 and April 2014.

ELIGIBILITY:
Inclusion Criteria:

* Patients having received a minimum of one platelet depletion procedure via the Spectra Optia system.
* Availability of complete blood count results prior to starting and after completing the platelet depletion procedure via the Spectra Optia system.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone platelet depletion via the Spectra Optia System and who were likely to have had blood disorders, such as essential thrombocythemia, a myeloproliferative disease, or reactive (secondary) thrombocytosis.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond P Goodrich, PhD, Study Director — VP, Scientific and Clinical Affairs; Chief Science Officer-BBT
Locations (2):
- Aarhus University Hospital, Aarhus, Denmark
- University of Pécs, Pécs, Hungary

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Who Received a Minimum of 1 PLTD Procedure u: Eligible subjects had received a minimum of 1 PLTD procedure using the Spectra Optia Apheresis System and had available pre- and post-procedure PLT counts.
Period: Overall Study
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Started | 12 (Data were collected from 20 PLTD procedures performed in 12 subjects)
Completed | 12 (Data were collected from 20 PLTD procedures performed in 12 subjects)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible subjects had received a minimum of 1 PLTD procedure using the Spectra Optia Apheresis System and had available pre- and post-procedure PLT counts.Data were collected from 20 PLTD procedures performed in 12 subjects, which constituted the Full and Safety Analysis Sets.
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years) | 64.3 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Region of Enrollment [Number; unit: participants]
  Denmark | 3
  Hungary | 9
Weight [Mean (Standard Deviation); unit: kg] | 63.6 (13.4)
Height [Mean (Standard Deviation); unit: cm] | 163.9 (9.2)
Total Blood Volume [Mean (Standard Deviation); unit: Liters] — Estimated by Nadler's formula for total blood volume of a human based on gender, height, and weight.
  Liters | 4.0 (0.7)
Diagnosis [Number; unit: pariticpants]
  Essential thrombocythaemia | 9
  Chronic myeloid leukaemia | 1
  Myelodysplastic/myeloproliferative neoplasm | 1
  Polycythaemia vera | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Platelet (PLT) Count in Patient Blood Following Apheresis Procedure
Description: (PLTpre - PLTpost) / PLTpre x 100%
Time Frame: on average this will be within 15 minutes after the end of the procedure
Population: Data were collected for 12 subjects who underwent a total of 20 PLTD procedures at 2 European sites.
Measure: Mean (Standard Deviation); unit: % change in PLT count in subject blood
Units Other Than Participants: procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number analyzed (procedures) | 20
% change in PLT count in subject blood | -58.2 (12.0)

2. Primary Outcome: Percent of Processed Platelets (PLT) Which Are Collected i.e. Collection Efficiency for Platelets Achieved by Spectra Optia.
Description: (PLT/µL product x product volume) / ((PLTpre + PLTpost) / 2) x total processed blood volume)
Time Frame: on average this will be within 15 minutes after the end of the procedure
Population: At Site 2, percent processed platelets could only be calculated for 1 procedure in Subject 214; no waste bag (depletion product) platelet counts were available for the other 9 procedures performed at Site 2.
Measure: Mean (Standard Deviation); unit: % of processed platelets
Units Other Than Participants: Procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 4
Number analyzed (Procedures) | 11
% of processed platelets | 67.8 (18.3)

3. Primary Outcome: Adverse Events
Time Frame: during the apheresis procedure (from the moment the patient is connected until he is disconnected from the device) and device or procedure related adverse events until discharge from Apheresis Unit (On average, half hour after end of procedure).
Population: Eligible subjects had received a minimum of 1 PLTD procedure using the Spectra Optia Apheresis System and had available pre- and post-procedure PLT counts.
Measure: Number; unit: Number of subjects with at least 1 AE
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number of subjects with at least 1 AE | 6

4. Other Pre Specified Outcome: Patient's Platelet Count Pre-depletion Procedure
Time Frame: Prior to each Spectra Optia Apheresis Procedure
Population: Data were collected for 12 subjects who underwent a total of 20 PLTD procedures at 2 European sites.
Measure: Mean (Standard Deviation); unit: cells x 10^3/L
Units Other Than Participants: procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number analyzed (procedures) | 20
cells x 10^3/L | 1740.7 (744.95)

5. Other Pre Specified Outcome: Patient's Platelet Count Post-depletion Procedure
Time Frame: Participants were followed for the duration of the procedure and an average of 2.5 hours after the procedure
Population: Data were collected for 12 subjects who underwent a total of 20 PLTD procedures at 2 European sites.
Measure: Mean (Standard Deviation); unit: cells x 10^3/L
Units Other Than Participants: procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number analyzed (procedures) | 20
cells x 10^3/L | 717.2 (336)

6. Other Pre Specified Outcome: Patients WBC Count Pre-depletion Procedure
Time Frame: Prior to each Spectra Optia Apheresis Procedure
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Units Other Than Participants: procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number analyzed (procedures) | 20
cells x 10^9/L | 15.9 (18.29)

7. Other Pre Specified Outcome: Patient's WBC Count Post-depletion Procedure
Time Frame: Participants were followed for the duration of the procedure and an average of 2.5 hours after the procedure
Population: Data were collected for 12 subjects who underwent a total of 20 PLTD procedures at 2 European sites.
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Units Other Than Participants: procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number analyzed (procedures) | 20
cells x 10^9/L | 8.4 (6.66)

8. Other Pre Specified Outcome: Whole Blood Processed (mL)
Description: Volume of patients blood processed during the apheresis procedure.
Time Frame: Post each Spectra Optia Apheresis Procedure
Population: Data were collected for 12 subjects who underwent a total of 20 PLTD procedures at 2 European sites.
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number analyzed (procedures) | 20
mL | 6652.3 (856.42)

9. Other Pre Specified Outcome: Average Inlet Flow Rate
Time Frame: Participants were followed for the duration of the procedure and an average of 2.5 hours after the procedure
Population: Data were collected for 12 subjects who underwent a total of 20 PLTD procedures at 2 European sites.
Measure: Mean (Standard Deviation); unit: mL/min
Units Other Than Participants: procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number analyzed (procedures) | 20
mL/min | 46.7 (8.45)

10. Other Pre Specified Outcome: Procedure Duration
Time Frame: Participants were followed for the duration of the procedure and an average of 2.5 hours after the procedure
Population: Data were collected for 12 subjects who underwent a total of 20 PLTD procedures at 2 European sites.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number analyzed (procedures) | 20
minutes | 144.5 (17.81)

11. Other Pre Specified Outcome: Waste Bag Volume
Time Frame: Post each Spectra Optia Apheresis Procedure
Population: Data were collected for 12 subjects who underwent a total of 20 PLTD procedures at 2 European sites.
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number analyzed (procedures) | 20
mL | 669.8 (248.48)

12. Other Pre Specified Outcome: Total Blood Volume (TBV) Processed
Description: The number of times the patient's total blood volume is processed during the apheresis procedure.
Time Frame: Post each Spectra Optia Apheresis Procedure
Population: Data were collected for 12 subjects who underwent a total of 20 PLTD procedures at 2 European sites.
Measure: Mean (Standard Deviation); unit: Number of TBVs processed
Units Other Than Participants: procedures
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Number analyzed (Participants) | 12
Number analyzed (procedures) | 20
Number of TBVs processed | 1.7 (0.25)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data (including serious adverse events [SAEs]) were collected from the time of the start of the PLTD procedure until discharge from the Apheresis Unit.
Description: Adverse events were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, and coded using the Medical Dictionary for Regulatory Activities (MedDRA®, Version 17.0).
Arm/Group | Subjects Who Received a Minimum of 1 PLTD Procedure u
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Who Received a Minimum of 1 PLTD Procedure u (N=12)
Anemia (Blood and lymphatic system disorders) | 3
Hypotension (Vascular disorders) | 3
Dizziness (Nervous system disorders) | 1
Malaise (General disorders) | 1
White blood cell count decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Site reserves the right to publish the results of its work on the Study. Study Site and the PI agree to submit copies of any manuscript/abstract proposed for publication to Sponsor at least 30 days in advance of the presentation. Sponsor may require the delay of publication for no longer than 90 days for the purpose of filing patent applications.